CLINICAL TRIAL: NCT06852196
Title: Time and Type Dependent Evaluation of Different Techniques for Correction of Cleft Maxillary Hypoplasia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abdullah Hashim Ahmed, Assistant lecturer of plastic surgery, Assiut University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Cleft Maxillary Hypoplasia
Record Dates: First submitted 2025-02-10; First posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Maxillary Hypoplasia; Cleft Lip Palate; Orthognathic Surgery
Keywords: cleft maxillary hypoplasia
MeSH Terms: conditions — Retrognathia | interventions — Osteogenesis, Distraction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- surgery first (Experimental): modern surgery-first orthognathic surgery approach (reduced treatment time, efficient tooth decompensation, and early improvement in facial esthetics),
  Interventions: Procedure: orthognathic surgery ,lefort 1,bsso ,DO; Procedure: distraction osteogenesis
- othodontics first (Experimental): orthodontics first then surgery
  Interventions: Procedure: orthognathic surgery ,lefort 1,bsso ,DO; Procedure: distraction osteogenesis

INTERVENTIONS:
Procedure: orthognathic surgery ,lefort 1,bsso ,DO — Le Fort I osteotomy is often used in the correction of dental occlusion and maxillary hypoplasia in cleft patients. In addition, the osteotomy may also improve patients' facial appearance and self-esteem
Procedure: distraction osteogenesis — Distraction osteogenesis is a surgical technique that uses body's own repairing mechanisms for optimal reconstruction of the tissues.

SUMMARY:
Maxillary hypoplasia in CLP deformities results from congenital reduction in midfacial growth and the effects of the surgical scar from CLP repair.Turvey et al. suggested that this disproportionate jaw growth is the biologic consequence of prior surgical intervention for closure of the soft tissues and is not related to the congenital cleft deformity, Midfacial hypoplasia is commonly treated by performing conventional Le Fort surgery to displace the maxilla anteriorly and stabilization afterward with rigid fixation along with orthodontics treatment. .

Midface hypoplasia cleft patient has the following characteristics: concave facial profile, inverted nasal tip, wide alar base, acute nasolabial angle, and excessive exposure of sclera. Intraoral findings are anterior and posterior crossbite, CLP, accentuated curve of Spee, Class III dental malocclusion, multiple missing teeth, oronasal communication, and residual cleft. Speech disturbances are also usually present due to velopharyngeal incompetency and oronasal communication.

ELIGIBILITY:
Inclusion Criteria:

* Cleft patients either cleft alveolus or cleft alveolus and palate.
* Surgically fit patients.
* Patients ready for orthognathic assessment undergoing either surgical or orthodontics correction.

Exclusion Criteria:

* Non- cleft cases .
* Previous correction.
* History of active infection or underlying disease such as hematologic disorders neoplasm, and immune deficiency.
* Patient refused to sign an informed consent.

Ages: 12 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 22 (Estimated)
Dates: Start 2025-02-21 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
CEPHALOMETRIC | 1 year
  MAXILLARY COMPONENT SNA (degrees) Sella to Nasion to point A angle normal angle is 82 degree plus or minus 3 degree

SECONDARY OUTCOMES:
facial canons | 1 year
  the rule of fifths, which divides the face in the transverse dimension into five equal parts by assuming that the intercanthal distance is equal to the nasal width and widths of the eyes, incorporates orbital and orbito-nasal canons
  and three equal lengths of the face (the forehead, the nose, and the mouth and chin), as well as the intercanthal distance being equal to the eye fissure length measurement are in cm